CLINICAL TRIAL: NCT05063474
Title: Microvascular Reactivity in People With Peripheral Artery Disease: a Pilot Study to Determine Reliability, Validity, and Sensitivity to Change
Brief Title: Microvascular Reactivity in Peripheral Artery Disease
Status: Terminated | Type: Observational
Why Stopped: Poor enrollment and lack of funding
Sponsor: Columbia University (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: AAAT5119; R01HS025198 (AHRQ)
Record Dates: First submitted 2021-09-09; First posted 2021-10-01 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Peripheral Artery Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PAD: Peripheral Artery Disease: People with Peripheral Artery Disease (PAD). No intervention given, observation and assessment only
  Interventions: Diagnostic Test: No Intervention-Clinical Assessments only
- PLL+PAD: People with Limb Loss and Peripheral Artery Disease: People with Lower-Limb Loss (PLL) and Peripheral Artery Disease (PAD) No intervention given, observation and assessment only
  Interventions: Diagnostic Test: No Intervention-Clinical Assessments only

INTERVENTIONS:
Diagnostic Test: No Intervention-Clinical Assessments only — No Intervention. Clinical Assessments include: vital signs, near infrared spectrometry, general leg strength, and 6-minute walking test.

SUMMARY:
Peripheral Artery Disease (PAD) is a major risk factor for lower limb amputation. Microvascular reactivity assessed with near-infrared spectrometry has been studied in people with PAD but not in people with limb loss (PLL) who have PAD. The purpose of this research is to explore whether near-infrared spectrometry measures can contribute to identifying people at risk for amputation. Specific aims include: 1) Determine the test-retest reliability of near-infrared spectrometry measures in people with peripheral artery disease with or without major unilateral amputation. 2) Determine construct validity of near-infrared spectrometry measures compared to 6-Minute Walk Test, and time to claudication onset; and self-reported prosthetic mobility in people with transtibial amputation.

This methodologic prospective study with repeated assessments and long term phone follow-up every year to identify any subjects that undergo revascularization or amputation will include 2 groups of subjects: a PAD group enrolled from an out-patient walking program, and a PLL+PAD group who receive no care but have their walking step counts monitored.

DETAILED DESCRIPTION:
Subjects: Subjects with peripheral artery disease (PAD) with or without lower limb amputation will be recruited from PAD rehabilitation programs or support groups for people with limb loss (PLL) in the Columbia University Irving Medical Center system and New York City metropolitan area. Equal numbers (n=10) will be assigned to the people with PAD group and the PLL plus PAD (PLL+PAD) group. All subjects will be 35-80 years old at risk for amputation as determined by meeting any of the following criteria. 1) People with peripheral artery disease diagnosed by ankle-brachial index (ABI) <0.9 or 1.4. 2) People who have a history of endovascular or surgical revascularization for critical ischemia, or 3) People with previous major or minor unilateral lower limb loss due to PAD, with or without diabetes. Once informed written consent has been obtained Assessment sessions will depend on group assignment.

The PLL+PAD group will attend 2 assessment sessions: initial and 1-month follow-up assessments only. The PLL+PAD group will receive no intervention. However, a monitor will be used to remotely assess their general walking activity. At the end of the initial assessment, PLL will have daily step count assessed with a StepWatch4 step activity monitor strapped just above the lateral prosthetic ankle. The average daily step count will be derived from the last full week of 24- hour/day data collection closest in time to the next assessment, at which time the StepWatch4 will be removed. Between sessions, subjects will be encouraged to continue their usual activities; no directions regarding exercise, physical activity, or walking will be given. Data from the two sessions will be used to determine test-retest reliability (Aim 1). Near infrared spectrometry measurement data from the 1st session will be used to determine associations with walking performance measures (Aim 2).

The PAD group will attend 3 assessment sessions: initial, 1-month, and 2-month follow-up assessments. The PAD group will already be enrolled in a PAD rehabilitation program-independent of this research program-that consists of 2-3 times per week 1-hour sessions. Sessions include progressive treadmill training for 30- minute-including rest breaks as needed-with inclination added if tolerated. Also included is 30-minutes of calf and hamstring stretching and general strengthening including free weights for the upper limbs, cuff weights for the lower limbs, and repeated sit-to-stand and step functional training. The rehabilitation program consists of 24 sessions over 2 months and the number of sessions attended will be counted. If subjects opt for an additional 1-month of training session, they will undergo a 3-month follow-up assessment. Repeated measures data from the PAD group will be used to determine effect size change of the primary outcome measures (Aim 3).

Measures: All subjects at each session will complete a questionnaire and undergo clinical assessments. Follow up calls every 6 months will be made to determine medical outcome.

Questionnaire data will include individual characteristics, medical history, and self-report claudication scale. General health perception will be assessed with SF-12.

Clinical assessment will occur at each session and include vital signs, ankle brachial index, near infrared spectrometry during strength and walking assessments. General lower extremity strength will be assessed with heel raises up to 25 repetitions and the 30-sec sit-to-stand. Walking performance will be assessed using the 6-Minute Walk Test using a standard 20m walkway with rests allowed as needed. Walking speed will be obtained from the first 20m. Clinical assessment of strength and walking are expected to be of moderate intensity.

Statistical analysis will include group descriptions, Intraclass Correlation Coefficients for test-retest reliability, and Pearson correlation coefficients for convergent or divergent validity between near infrared spectrometry and clinical outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* People of any sex or race/culture
* Clinical diagnosed of peripheral artery disease
* People with or without diabetes
* People with or without past endovascular or vascular procedures for peripheral artery disease within the past year
* People who have unilateral minor or major lower limb amputation

Exclusion Criteria:

* People who cannot communicate in English
* People judged unable to participate due to cognitive limitation or medical instability
* People who cannot walk independently 50 feet, with or without walking aid

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with peripheral artery disease with or without lower limb amputation will be recruited from peripheral artery disease (PAD) rehabilitation programs or support groups for people with limb loss (PLL) in the Columbia University Irving Medical Center system and New York City metropolitan area. Equal numbers (n=10) will be assigned to the people with PAD group and the PLL plus PAD (PLL+PAD) group.
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2021-11-09 (Actual); Primary Completion 2023-04-24 (Actual); Study Completion 2023-04-24 (Actual)

PRIMARY OUTCOMES:
Microvascular Reactivity | Monthly: from initial assessment each month for up to 2 months.
  Near Infrared Spectrometry

SECONDARY OUTCOMES:
6-Minute Walk Test | Monthly: from initial assessment each month for up to 2 months.
  Distance and speed
Claudication | Monthly: from initial assessment each month for up to 2 months.
  Time to onset and severity
General Lower-Limb Strength | Monthly: from initial assessment each month for up to 2 months.
  30s Sit-to-Stand test
Calf muscle strength | Monthly: from initial assessment each month for up to 2 months.
  Repetitive heel raises (up to 25 max)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher K Wong, PhD, PT, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barnes JA, Eid MA, Creager MA, Goodney PP. Epidemiology and Risk of Amputation in Patients With Diabetes Mellitus and Peripheral Artery Disease. Arterioscler Thromb Vasc Biol. 2020 Aug;40(8):1808-1817. doi: 10.1161/ATVBAHA.120.314595. Epub 2020 Jun 25. PMID 32580632
- [Background] Vieira de Oliveira G, Soares RN, Volino-Souza M, Murias JM, Alvares TS. The association between near-infrared spectroscopy assessment of microvascular reactivity and flow-mediated dilation is disrupted in individuals at high risk for cardiovascular disease. Microcirculation. 2019 Oct;26(7):e12556. doi: 10.1111/micc.12556. Epub 2019 Jun 2. PMID 31077636
- [Background] Duscha BD, Piner LW, Patel MP, Crawford LE, Jones WS, Patel MR, Kraus WE. Effects of a 12-Week mHealth Program on FunctionalCapacity and Physical Activity in Patients With PeripheralArtery Disease. Am J Cardiol. 2018 Sep 1;122(5):879-884. doi: 10.1016/j.amjcard.2018.05.018. Epub 2018 Jun 2. PMID 30049464
- [Background] Behroozian A, Beckman JA. Microvascular Disease Increases Amputation in Patients With Peripheral Artery Disease. Arterioscler Thromb Vasc Biol. 2020 Mar;40(3):534-540. doi: 10.1161/ATVBAHA.119.312859. Epub 2020 Feb 20. PMID 32075418
- [Background] Criqui MH, Aboyans V. Epidemiology of peripheral artery disease. Circ Res. 2015 Apr 24;116(9):1509-26. doi: 10.1161/CIRCRESAHA.116.303849. PMID 25908725
- [Background] Olin JW, White CJ, Armstrong EJ, Kadian-Dodov D, Hiatt WR. Peripheral Artery Disease: Evolving Role of Exercise, Medical Therapy, and Endovascular Options. J Am Coll Cardiol. 2016 Mar 22;67(11):1338-57. doi: 10.1016/j.jacc.2015.12.049. PMID 26988957
- [Background] Jones S, Chiesa ST, Chaturvedi N, Hughes AD. Recent developments in near-infrared spectroscopy (NIRS) for the assessment of local skeletal muscle microvascular function and capacity to utilise oxygen. Artery Res. 2016 Dec;16:25-33. doi: 10.1016/j.artres.2016.09.001. PMID 27942271